CLINICAL TRIAL: NCT00023842
Title: A Randomized Phase II Trial of Sequential Chemo-Immunotherapy Versus Immunotherapy Alone in Carcinoma in Situ of the Urinary Bladder
Brief Title: BCG With or Without Mitomycin in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30993; EORTC-30993; AURO-EORTC-30993; FINNBLADDER-EORTC-30993; GAUO-EORTC-30993; SEUG-EORTC-30993; UKCCCR-EORTC-30993; NCRI-EORTC-30993
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; recurrent bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; Mitomycin; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: BCG vaccine
Drug: mitomycin C
Procedure: adjuvant therapy
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies such as BCG use different ways to stimulate the immune system and stop tumor cells from growing. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with biological therapy may kill more tumor cells. It is not yet known if BCG is more effective with or without mitomycin.

PURPOSE: Randomized phase II trial to compare the effectiveness of BCG plus mitomycin with that of BCG alone in treating patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the complete response rate of patients with carcinoma in situ of the bladder treated with adjuvant intravesical BCG with or without intravesical mitomycin following transurethral resection.
* Compare the disease-free interval and type of recurrence after complete response in patients treated with these regimens.
* Compare the side effects of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to one of two treatment arms.

Arm I:

* Induction therapy: Patients receive intravesical mitomycin over 1 hour once weekly on weeks 1-6 and intravesical BCG once weekly on weeks 7-12. Patients with visible lesions or disease recurrence or progression undergo transurethral resection (TUR) during weeks 16-18 and receive one additional course of intravesical therapy.
* Maintenance therapy:Patients with a complete response after either course of induction therapy proceed to maintenance therapy comprising intravesical mitomycin once on week 1 and intravesical BCG once weekly on weeks 2 and 3. Maintenance therapy repeats every 6 months through year 3.

Arm II:

* Induction therapy:Patients receive intravesical BCG once weekly on weeks 1-6 and 10-12. Patients with visible lesions or disease recurrence or progression undergo transurethral resection (TUR) during weeks 16-18 and receive one additional course of intravesical therapy.
* Maintenance therapy: Patients with a complete response after either course of induction therapy receive maintenance therapy comprising intravesical BCG once weekly on weeks 1-3. Maintenance therapy repeats every 6 months through year 3.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 84-126 patients (42-63 per treatment arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma in situ (CIS) of the bladder with urinary cytology

  * Primary CIS (no prior history of CIS, papillary, or solid transitional cell carcinoma [TCC] of the bladder and no concurrent papillary or solid TCC) OR
  * Secondary CIS (detected after complete resection of superficial Ta/T1 TCC of the bladder) OR
  * Concurrent CIS (in the presence of superficial primary or recurrent Ta/T1 TCC of the bladder)
* No more than 28 days since prior transurethral resection (TUR) of all visible lesions
* No muscle involvement
* No prior or concurrent upper urinary tract tumors
* No urethral strictures that would prevent endoscopic procedures and repeated catheterization
* No upper urinary tract disease (e.g., vesico-ureteral reflux or massive stones) that would make multiple transurethral procedures risky

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No active tuberculosis (highly positive skin tests allowed if no active disease)
* No disease that would preclude general anesthesia
* No active intractable or uncontrollable infection
* No other prior or concurrent malignancy except cured basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior BCG

Chemotherapy:

* More than 3 months since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the pelvis

Surgery:

* See Disease Characteristics

Other:

* More than 3 months since prior intravesical cytostatic agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2001-06; Primary Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo V. Bono, MD, Study Chair — Ospedale di Circolo e Fondazione Macchi
Locations (16):
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
- Italy (3):
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Universita Degli Studi Di Pisa, Pisa
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- Hospital Desterro, Amadora, Portugal
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)
- United Kingdom (2):
  - Bristol Royal Infirmary, Bristol, England
  - University of Wales College of Medicine, Cardiff, Wales

REFERENCES:
- [Result] Oosterlinck W, Kirkali Z, Sylvester R, da Silva FC, Busch C, Algaba F, Collette S, Bono A. Sequential intravesical chemoimmunotherapy with mitomycin C and bacillus Calmette-Guerin and with bacillus Calmette-Guerin alone in patients with carcinoma in situ of the urinary bladder: results of an EORTC genito-urinary group randomized phase 2 trial (30993). Eur Urol. 2011 Mar;59(3):438-46. doi: 10.1016/j.eururo.2010.11.038. Epub 2010 Dec 7. PMID 21156335